CLINICAL TRIAL: NCT03167645
Title: Does Perioperative Substitution of Albumin Deficiency Reduce Postoperative Complications?
Brief Title: SUbstition of PERioperative Albumin Deficiency Disorders
Acronym: SUPERADD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUPERADD; 2016-001313-24 (EudraCT Number)
Record Dates: First submitted 2016-10-18; First posted 2017-05-30 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hypoalbuminemia
MeSH Terms: conditions — Hypoalbuminemia | interventions — Serum Albumin, Human; Albumins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human albumin (Experimental): Substitution of human albumin until serum albumin >30g/l; dosage: (30 g/l - serum albumin [g/l] ) x 0,04 l/kg x body weight [kg] x 2
  Interventions: Drug: Human albumin
- Control (No Intervention): Standard clinical care

INTERVENTIONS:
Drug: Human albumin — Substitution according to pre-specified dosage
  Other Names: Human-Albumin 20 % Behring, salzarm
  Arms: Human albumin

SUMMARY:
Aim of this study is to reduce postoperative complications (assessed by POMS-Score and graded by Clavien-Dindo-Score) by substitution of perioperative hypoalbuminaemia in high-risk patients or patients undergoing high risk surgery.

DETAILED DESCRIPTION:
Perioperative hypoalbuminaemia is a common condition in high risk surgery and in high risk patients. It is associated with increased morbidity and mortality. Although many studies investigated albumin substitution in critically ill patients there is still no clear recommendation for its use over any other colloid. Except for some smaller studies especially in the setting of cardiac surgery the effect of perioperative albumin substitution has not been studied yet.

This study is designed to investigate the effect of perioperative albumin substitution in high risk patients or patients undergoing high risk surgery on postoperative complications assessed by the POMS-Score and graded according to severity by the Clavien-Dindo-Score.

Patients eligible for the study are informed in detail during the pre-medication visit and written informed consent will be obtained. Additionally the Quality of Recovery 9 Score (QoR-9) will be determined. During induction of anesthesia blood is taken from every patient and the serum albumin level is determined. In case albumin is greater than 30 g/l albumin levels are controlled every 3 hours and one last time on admission to the postoperative anaesthesia care unit (PACU). Should the albumin level do not fall below 30 g/l over the whole period the patient is not randomized.

Patients with albumin ≤30g/l will be randomized using a web-based computer-generated randomization list into one of two groups:

Group human albumin (HA):

In this group hypoalbuminaemia is treated with infusion of human albumin until serum albumin is greater than 30g/l. To verify success of the therapy, serum albumin levels are controlled every 3 hours during surgery, on admission to the PACU and if necessary again in the PACU.

Group control:

In this group patients are treated according to standard clinical care. To compare the effect of albumin substitution serum albumin is measured every 3 hours from beginning of anesthesia until discharge from the PACU.

In both groups patients will be discharged from the PACU when the patient is rated fit for discharge by the attending anesthetist and albumin level is >30g/l in the HA group.

A blinded investigator assesses the patients postoperative complications. He visits the patient on day 3, 5, 8 and 15 after surgery and determines the POMS-score (see reference: Grocott MP). If a complication is detected the assessor grades the complication according to its severity with the Clavien-Dindo-Score (see reference: Clavien PA). Additionally serum albumin and creatinine levels will be determined in routine blood tests. The patients QoR-9, the Charlson Comorbidity Score, the Preoperative Score to Predict Postoperative Mortality (POSPOM) and other secondary outcome (see Outcome Measures section) parameters will be obtained.

6 Month after surgery the patient or next of kin will be contacted in order to determine 6-month mortality and the QoR-9 score.

Postulating an incidence of complications (graded Clavien-Dindo-Score 2 or higher) of 52% in group control and a reduced incidence of 38% in group HA results in a total number of 400 patients (chi-square-test, α = 0,048, power 80%). As the actual incidence is unknown but has a significant impact on the number needed per group, an interims analysis will be performed after 100 included patients. Is the difference of the incidence of postoperative complications between the two groups significant with an α < 0,002 the study will be finished. Otherwise, the sample size needed per group will be corrected assuming a relative risk reduction of 25% (52% vs. 38%), an α = 0,048, a two-tailed test and a power of 80%.

The blinded and independent interims analysis after 100 patients revealed a corrected sample size of 300 patients per group (total 600 patients).

ELIGIBILITY:
Inclusion Criteria:

* age: 18 years or older
* written informed consent
* ASA state 3 and 4 OR
* elective high risk surgery (open aortic surgery, open leg revascularization, thrombectomy, oesophagectomy, pancreatic surgery, cystectomy, liver surgery, change of knee- or hip-prothesis, amputation)

Exclusion Criteria:

* emergency surgery
* severe liver cirrhosis (child pugh C)
* need for dialysis
* patients already included in SUPERADD
* patients with a legal representative
* contraindications for human albumin: hypersensitivity for human albumin or any substance included in the preparation
* pregnancy
* breastfeeding women
* ASA state 5
* BMI > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Postoperative complications assessed with POMS- and graded with Clavien-Dindo-Score | 15 days
  Postoperative complications will be detected using the POMS score. The severity of the complications will be graded with the Clavien-Dindo-Score. A complication will be regarded as clinical relevant when it is graded Clavien-Dindo-Score 2 or higher on at least one of the four days examined.

SECONDARY OUTCOMES:
Length of hospital stay | until discharge from hospital, up to 6 month
Length of stay in postoperative anaesthesia care unit | until discharge from postoperative anaesthesia care unit, up to 24 hours
Length of stay in intensive care unit | until discharge from intensive care unit, up to 1 month
Long term mortality (6 month) | 6 month
Short term mortality (hospital mortality) | until discharge from hospital, up to 6 month
Acute kidney injury | until discharge from hospital, up to 6 month
  Incidence according to AKIN score (at least AKIN 1)
Quality of Recovery 9 Score | 6 month after surgery
  Assessed preoperatively and on day 1 and 3 an 6 month after surgery
Amount of volume infused | until discharge from postoperative anaesthesia care unit, up to 24 hours
  Amount of infusion of ringer's acetate and gelafundin
Dosage of catecholamines | until discharge from postoperative anaesthesia care unit, up to 24 hours
  Intra- and postoperative dosage of catecholamines
Number of red packed cells transfused | until discharge from postoperative anaesthesia care unit, up to 24 hours
Number of platelet concentrates transfused | until discharge from postoperative anaesthesia care unit, up to 24 hours
Amount of coagulation factors infused | until discharge from postoperative anaesthesia care unit, up to 24 hours
  Amount of PPSB and fibrinogen
Intra- and postoperative Hypotension | until discharge from postoperative anaesthesia care unit, up to 24 hours
  Decrease of more than 30% compared to value before induction
Incidence of pulmonal venous congestion | until discharge from postoperative anaesthesia care unit, up to 24 hours
  Incidence of pulmonal venous congestion assessed using chest x-ray
Therapy with diuretics | until discharge from hospital, up to 6 month
  New onset or extension of diuretic treatment
Efficacy of albumin treatment | until discharge from hospital, up to 6 month
  Efficacy of albumin treatment in order to increase serum albumin and colloid osmotic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, MD, Principal Investigator — Klinikum rechts der Isar, Technical University Munich, Dept. of Anesthesiology
Locations (1):
- Klinikum rechts der Isar Dept. of Anesthesiology, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clavien PA, Sanabria JR, Strasberg SM. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Surgery. 1992 May;111(5):518-26. PMID 1598671
- [Background] Grocott MP, Browne JP, Van der Meulen J, Matejowsky C, Mutch M, Hamilton MA, Levett DZ, Emberton M, Haddad FS, Mythen MG. The Postoperative Morbidity Survey was validated and used to describe morbidity after major surgery. J Clin Epidemiol. 2007 Sep;60(9):919-28. doi: 10.1016/j.jclinepi.2006.12.003. Epub 2007 May 7. PMID 17689808
- [Derived] Schaller SJ, Fuest K, Ulm B, Schmid S, Bubb C, von Eisenhart-Rothe R, Friess H, Kirchhoff C, Stadlbauer T, Luppa P, Blobner M, Jungwirth B. Substitution of perioperative albumin deficiency disorders (SuperAdd) in adults undergoing vascular, abdominal, trauma, or orthopedic surgery: protocol for a randomized controlled trial. Trials. 2020 Aug 18;21(1):726. doi: 10.1186/s13063-020-04626-2. PMID 32811539